CLINICAL TRIAL: NCT07383155
Title: Bivalirudin Versus Heparin During PCI in High Bleeding Risk Patients With Acute Coronary Syndromes
Acronym: BRIGHT-HBR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Professor, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRIGHT-HBR; 2025ZD0546400 (Other Grant/Funding Number: Noncommunicable Chronic Diseases-National Science and Technology Major Project of China)
Record Dates: First submitted 2026-01-24; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Percutaneous Coronary Intervention; High Bleeding Risk; Acute Coronary Syndromes; Anticoagulant Therapy
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Bivalirudin
  Interventions: Drug: Anticoagulant Therapy
- Group 2 (Active Comparator): Unfractionated heparin monotherapy
  Interventions: Drug: Anticoagulant Therapy

INTERVENTIONS:
Drug: Anticoagulant Therapy — The optimal parenteral anticoagulant during percutaneous coronary intervention (PCI) in high bleeding risk (HBR) patients with acute coronary syndromes (ACS)

SUMMARY:
Background. Randomized data on the optimal parenteral anticoagulant during percutaneous coronary intervention (PCI) in high bleeding risk (HBR) patients with acute coronary syndromes (ACS) are lacking.

Methods. BRIGHT-HBR is an investigator-sponsored, open-label, randomized controlled trial comparing bivalirudin vs. unfractionated heparin (UFH) monotherapy in HBR patients with ACS undergoing PCI. A total of 5270 HBR patients with a non-ST-elevation acute coronary syndrome (NSTE-ACS) or recent stabilized ST-segment elevation myocardial infarction (STEMI, ≥48 hours after symptom onset) will be randomized 1:1 to bivalirudin or UFH at 70 sites in China. HBR is defined by the Academic Research Consortium (ARC)-HBR criteria. The primary composite endpoint is net adverse clinical events (NACE) at 30 days, the composite of all-cause death, myocardial infarction, stroke, urgent target-vessel revascularization, or BARC types 2, 3 or 5 bleeding, and the major secondary endpoint is BARC types 2, 3 or 5 bleeding. The study is powered to demonstrate that bivalirudin is superior to UFH monotherapy for NACE in ACS patients with HRB at 30 days after PCI.

Conclusions. The BRIGHT-HBR randomized trial aims to provide evidence on whether bivalirudin reduces the incidence of NACE and clinically relevant bleeding compared with UFH monotherapy in patients with ACS who are at HBR undergoing PCI.

DETAILED DESCRIPTION:
Study design BRIGHT-HBR is an investigator-sponsored, prospective, multicenter, open-label, active-controlled randomized trial. A total of 5,270 patients with NSTE-ACS and stabilized recent STEMI who are at HBR and are undergoing PCI with radial artery access will be enrolled at 70 sites in China. Patients are randomized 1:1 to two arms: bivalirudin vs. UFH monotherapy, with GPI reserved for bailout use in each group. The trial is powered to demonstrate the superiority of bivalirudin compared with UFH in reducing the 30-day rate of net adverse clinical events (NACE), the composite of all-cause death, MI, stroke, urgent target-vessel revascularization, or bleeding according to the Bleeding Academic Research Consortium (BARC) types 2, 3 or 5 criteria.

Randomization and study treatment Before diagnostic angiography, eligible patients will be randomly assigned in a 1:1 ratio to procedural anticoagulation with bivalirudin or UFH monotherapy. Allocation to treatment will be provided by an interactive web response system in randomly permuted block sizes of 4 or 6, with stratification according to the participating center, which is incorporated within an electronic data capture system.

In the UFH monotherapy group, an intravenous UFH bolus of 70 U/kg will be administered. The ACT will be measured 5 minutes after the first administration, and if the ACT is <250 seconds (Hemotec assay), an additional intravenous bolus of 1000 U UFH will be administered, to ensure the re-checked ACT is ≥250 seconds prior to PCI.

In the bivalirudin group, an intravenous bolus dose of bivalirudin 0.75 mg/kg will be administered, followed by an intravenous infusion of 1.75 mg/(kg·h). The infusion dose (but not the bolus) is adjusted for renal insufficiency. The estimated glomerular filtration rate (eGFR) will be calculated by the formula: 186 × (serum creatinine [mg/dL])-1.154 × (age)-0.203 × (0.742 if female). For patients with moderate renal impairment (eGFR 30-59 ml/(min·1.73m2), the intravenous infusion dose is unchanged; for patients with severe renal impairment (eGFR <30 ml/(min·1.73m2), the intravenous infusion dose is reduced to 1.0 mg/(kg·h); for patients undergoing dialysis, the intravenous infusion dose is reduced to 0.25 mg/(kg·h). The ACT will be monitored 5 minutes after the first bivalirudin bolus administration, and if the ACT is <250 seconds (Hemotec assay), an additional intravenous bolus of 0.3 mg/kg of bivalirudin will be administered to ensure the re-checked ACT is ≥250 seconds prior to PCI. The intravenous bivalirudin infusion is discontinued immediately after PCI.

The PCI procedure is performed using standard techniques. Radial artery access is strongly recommended. PCI is recommended for vessels with a visually assessed coronary artery diameter ≥2.5 mm with stenosis ≥70% or fractional flow reserve (FFR) <0.80 or ulcerated plaques. Complete revascularization is recommended if it may be safely achieved. PCI of chronic total occlusions (CTO) that are well-collateralized and supply viable myocardium is recommended if, in the opinion of an experienced CTO operator, there is a high likelihood of PCI success without complications or excessive contrast use. Drug-eluting stents should be used absent contraindications. Declaration of the target vessels will be made before PCI. A planned staged procedure in patients with complex or multivessel disease may be completed within 45 days and will not be considered an endpoint event. The intent to stage must be declared and documented at the end of the first procedure. The anticoagulation regimen during the planned staged procedure must be identical with that of the initial procedure. Any unplanned treatment, or a planned reintervention after 45 days will be considered an endpoint event.

Routine administration of a GPI during the procedure is prohibited. The use of intravenous or intracoronary tirofiban (the most widely used GPI in China) is restricted to specific procedural complications, including target vessel slow flow or no-reflow, refractory thrombus, or other thrombotic complications during PCI that cannot otherwise be effectively treated. When indicated, intravenous tirofiban should be initiated with a bolus infusion of 10-25 μg/kg (administered over >5 minutes), followed by a continuous maintenance infusion of 0.15 μg/(kg·min) for up to 18 hours. For patients with an eGFR <60 mL/min, the maintenance dose should be reduced to 0.075 μg/(kg·min). Alternatively, an intracoronary bolus dose of 500-750 μg may be used, with repeat injections permitted at intervals of 3-5 minutes. The cumulative intracoronary dose should not exceed 1500-2250 μg. Other procedural medications are provided per standard of care.

Prior to the procedure the patient should be treated with aspirin and a standard loading dose followed by a daily dose of either ticagrelor or clopidogrel (ticagrelor strongly preferred). Dual antiplatelet therapy should be continued post-PCI per local standard of care and societal guidelines. Other chronic medications are administered per local standard of care.

Follow-up Clinical follow-up will be scheduled at 1, 3, 6, and 12 months via telephone or clinic visit after randomization. Throughout the study period, patients will be monitored for the occurrence of the following clinical events: death, MI, stroke, any repeat revascularization, and any bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical evidence of NSTE-ACS or recent stabilized STEMI (≥48 hours after symptom onset) undergoing PCI
* The patient meets the ARC criteria for HBR (≥1 major criterion or ≥2 minor criteria)
* The patient or legal representative has been fully informed and written informed consent has been obtained

Exclusion Criteria:

* STEMI patients within 48 hours of symptom onset
* CABG or PCI within the prior 6 months, including for the present clinical syndrome
* Cardiogenic shock
* Coronary artery disease unsuitable for revascularization or requiring CABG
* Confirmed or suspected aortic dissection
* Treatment with a glycoprotein IIb/IIIa inhibitor within 2 hours prior to the PCI (use of intravenous heparin prior to or at the time of randomization is acceptable)
* Allergy to UFH, bivalirudin, aspirin, clopidogrel, ticagrelor, or contrast agents that cannot be adequately pre-medicated, or any prior anaphylaxis to these agents
* Any non-cardiac conditions with an expected life expectancy of ≤12 months
* Patients deemed by the investigator to be clinically unsuitable for coronary angiography and PCI, or who are unlikely to be able to comply with the protocol requirements, including medication adherence and follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5270 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical events (NACE) at 30 days | 30 days post PCI
  The composite of all-cause death, MI, stroke, urgent target-vessel revascularization, or BARC types 2, 3 or 5 bleeding

SECONDARY OUTCOMES:
BARC types 2, 3 or 5 bleeding at 30 days | 30 days post PCI
NACE at 12 months | 1 year post PCI
Each individual component of NACE at 30 days and 12 months | 30 days and 1 year post PCI
Major adverse cardiac and cerebral events (MACCE) at 30 days and 12 months | 30 days and 1 year post PCI
  Composite of all-cause death, MI, stroke, or urgent target-vessel revascularization
BARC types 1, 2, 3, or 5 bleeding at 30 days and 12 months | 30 days and 1 year post PCI
BARC types 3 or 5 bleeding at 30 days and 12 months | 30 days and 1 year post PCI
Definite/probable stent thrombosis at 30 days and 12 months | 30 days and 1 year post PCI

IPD SHARING:
Plan to Share IPD: Undecided